CLINICAL TRIAL: NCT05018559
Title: Physical Activity-related Health Competence in Apprenticeship and Vocational Education
Acronym: PArC-AVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Head of the Department of Sport Science and Sport, University of Erlangen-Nürnberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PArC-AVE
Record Dates: First submitted 2021-08-12; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Health Behavior
Keywords: physical activity promotion
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group nursing care (Experimental): Participants receive a co-created physical activity intervention called BuG lesson (German: 'Bewegt und Gesund'-Stunde; English: PA and health lesson).
  Interventions: Behavioral: BuG lesson
- Control group nursing care (No Intervention): Participants do not receive any treatment in addition to their vocational education and training curriculum.
- Intervention group automotive mechatronics (Experimental): Participants receive a co-created physical activity intervention called tutoring system.
  Interventions: Behavioral: Tutoring system
- Control group automotive mechatronics (No Intervention): Participants do not receive any treatment in addition to their vocational education and training curriculum.

INTERVENTIONS:
Behavioral: BuG lesson — Participants of the intervention group in nursing care received a co-created setting-specific intervention to promote physical activity called BuG lesson. The BuG lesson comprises a weekly 90-minute lesson for apprentices of nursing care during regular school hours, covering physical activity and health in theory and practice. Previously, the nursing teachers voluntarily underwent a qualification process as physical activity instructors, enabling them to conduct the BuG lessons independently.
  Arms: Intervention group nursing care
Behavioral: Tutoring system — Participants of the intervention group in automotive mechatronics received a co-created setting-specific intervention to promote physical activity called tutoring system. In the tutoring system, automotive mechatronics apprentices act as physical activity promotors for their fellow apprentices. In the sense of a peer-to-peer approach, apprentices voluntarily participate in a workshop to be qualified as tutors. Subsequently, the tutoring system takes place every two weeks for about ten to fifteen minutes during regular working hours, allowing the tutors to discuss the issues of physical activity and health among their peers.
  Arms: Intervention group automotive mechatronics

SUMMARY:
Although the health-promoting effects of physical activity are well known and apprentices often possess an insufficient amount of physical activity, there is a lack of interventions promoting physical activity in vocational education and training. Against this background, the PArC-AVE project uses a co-creation approach to develop and implement physical activity-promoting interventions tailored to the needs of the target group and the given setting in two vocational education and training institutions. The purpose of this study is to evaluate the effectiveness of the co-created interventions in vocational education and training, namely the BuG lesson in nursing care and the tutoring system in automotive mechatronics. Therefore, the investigators conducted two non-randomized controlled trials from October 2018 to September 2019.

ELIGIBILITY:
Inclusion Criteria:

* First-year apprentices from the automotive mechatronics and nursing care sectors

Exclusion Criteria:

* /

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Changes in self-reported physical activity: BSA questionnaire | Baseline and 6 to 9 months
  The Physical Activity, Exercise, and Sport Questionnaire (Bewegungs- und Sportaktivität Fragebogen; BSA-F) is a German questionnaire that assesses the amount of physical activity during the last four weeks. It differentiates between leisure-time/transportation activities (physical activity score) and sport-/exercise-related activities (sports score). Participants are required to report the frequency and duration of activities executed during the last four weeks. Minutes of leisure-time physical activity per week and sport-/exercise-related activity per week are calculated to get the physical activity and the sports score. Both scores can be combined to receive the overall volume of physical activity completed during leisure-time/transportation and sport-/exercise-related activities.
Changes in physical activity-related health competence: BGK Questionnaire | Baseline and 6 to 9 months
  This will be measured by the German version of the Physical Activity-Related Health Competence questionnaire. The questionnaire consists of 44 total items that measure three sub-competencies necessary for a health-promoting physical activity behavior: movement competence (20 items; min = 0, max = 17.6), control competence (10 items; min = 0, max = 10.8), physical activity-related self-regulation competence (14 items; min = 0, max = 14.8). Higher scores indicate higher competencies.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Principal Investigator — Friedrich-Alexander-University Erlangen-Nürnberg
Locations (1):
- Friedrich-Alexander-University Erlangen-Nürnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No
The datasets generated for this study are available from the corresponding author upon request.

REFERENCES:
- [Derived] Grune E, Popp J, Carl J, Semrau J, Pfeifer K. Examining the sustainability and effectiveness of co-created physical activity interventions in vocational education and training: a multimethod evaluation. BMC Public Health. 2022 Apr 15;22(1):765. doi: 10.1186/s12889-022-13133-9. PMID 35428289